CLINICAL TRIAL: NCT02525718
Title: Does Selective Intraoperative Administration of Local Anesthesia in Breast Reconstruction Reduce Postoperative Pain and Opioid Requirement?: A Prospective Double-Blinded Randomized Controlled Trial
Brief Title: Selective Intraoperative Administration of Local Anesthesia in Breast Reconstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mohammed Alghoul, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00200903
Record Dates: First submitted 2015-07-06; First posted 2015-08-17 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Breast Reconstruction; Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sodium Chloride; Bupivacaine; Epinephrine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be randomly selected to receive saline (placebo), administered to the breast area to cover the intercostal nerves supplying the breast tissue during surgery.
  Interventions: Drug: Saline
- 0.25 % bupivacaine w/ epinephrine & 4mg dexamethasone (Active Comparator): Subjects will be randomly selected to receive selective block with a local anesthetic solution containing 0.25 % bupivacaine (2.5 mg/ml) with 1:100,000 epinephrine and 4 mg dexamethasone. The injection will be performed in certain locations of the breast area to cover the intercostal nerves supplying the breast tissue.
  Subjects will be randomly selected to receive the local anesthetic solution containing 0.25 % bupivacaine (2.5 mg/ml) with 1:100,000 epinephrine and 4 mg dexamethasoneadministered to the breast area to cover the intercostal nerves supplying the breast tissue during surgery.
  Interventions: Drug: 0.25 % bupivacaine (2.5 mg/ml) w/ 1:100,000 epinephrine & 4 mg dexamethasone

INTERVENTIONS:
Drug: Saline — If randomized to this arm, subjects will receive an intraoperative injection of saline. (2.5 mg/ml)
  Other Names: Sodium Chloride 0.9%
  Arms: Placebo
Drug: 0.25 % bupivacaine (2.5 mg/ml) w/ 1:100,000 epinephrine & 4 mg dexamethasone — If randomized to this arm, subjects will receive a selective block with a local anesthetic solution containing 0.25 % bupivacaine.
  (2.5 mg/ml) with 1:100,000 epinephrine and 4 mg dexamethasone intraoperatively.
  Other Names: Bupivacaine
  Arms: 0.25 % bupivacaine w/ epinephrine & 4mg dexamethasone

SUMMARY:
Subjects are being asked to participate in this study because they will be undergoing unilateral (one) or bilateral (two) mastectomy surgery with immediate reconstruction involving insertion of a tissue expander.

DETAILED DESCRIPTION:
One in eight women will develop breast cancer in her lifetime, and many of these women undergo mastectomy followed by breast reconstruction by insertion of a tissue expander below the pectoralis major muscle. Women undergoing breast reconstruction have been shown to have a significantly higher level of acute postoperative pain and postoperative narcotic requirement compared to women who undergo mastectomy alone without reconstruction. In addition to the inherently worthwhile end of providing patient comfort in the immediate postoperative period, decreased narcotic use carries with it the potential benefit of decreasing the incidence of other adverse effects such as nausea, vomiting, allergic reaction, and respiratory depression.

Importantly, the intensity of pain in the immediate postoperative period has been implicated as an important factor predisposing patients to the development of chronic postoperative pain. Chronic pain following mastectomy is a significant and disabling problem, affecting up to 49% of patients in some series. Though breast reconstruction has been shown not to be an independent predictor of the development of chronic breast pain, improved control of acute pain in the immediate postoperative period carries significant promise in decreasing the incidence of this disabling condition for all breast cancer survivors treated with mastectomy. In addition, improving management of acute postoperative pain can shorten hospital stay, expedite return to daily normal activities and increase patient satisfaction.

A variety of other adjuncts for pain control have been attempted in studies of variable methodological rigor, including injection of botulinum toxin into the pectoralis muscle, indwelling pain catheters, paravertebral blocks under ultrasound guidance, or simple irrigation of the general area of dissection during breast surgery with a solution containing local anesthestic. While each of these adjuncts has demonstrated some success, none has been widely adopted. Problems with these methods include cost, risk of adverse events, as well as anatomically incomplete or non-selective application.

During mastectomy all breast tissue is removed, leaving the patient with denervated skin flaps. For breast reconstruction, a tissue expander is placed in a subpectoral pocket dissected between the pectoralis major and minor muscles. At the end of the procedure the pectoralis major muscle is placed under variable degree of tension depending on the amount of fluid placed inside the expander. This muscle stretch believed to be at least partially responsible for postoperative pain. In addition cut nerve endings in the superficial fascia likely contribute as well. The anatomy of nerves supplying the breast and involved muscles are well-described in rigorous cadaver studies.

In this study we hypothesize that performing a block of the intercostal nerves responsible for innervating the breast tissue and skin and the pectoral nerves innervating the pectoralis major muscle should optimize immediate postoperative pain control in this patient population. Of adjuncts described in the literature, paravertebral blocks are the most anatomically targeted, but drawbacks include the need for a separate procedure preoperatively while the patient is awake by an anesthesiologist with facility performing these blocks as well as the risk of pneumothorax. Advantages of our proposed method include lack of pain as the patient is asleep, easy and speed of application, a decreased risk of pneumothorax as the injections are under direct visualization, as well as a decrease in cost and improved efficiency as the only a single provider (i.e. the operative surgeon) is required. Precedent for our technique has been described in the context of breast augmentation and breast lift, with a favorable safety profile and providing adequate analgesia to perform these procedures without the use of a general anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo mastectomy surgery with immediate reconstruction involving insertion of a tissue expander performed by the principal investigator beginning from the time of study approval until study enrollment is complete.

Exclusion Criteria:

* Patients under the age of 18, or over the age of 79
* Allergy to local anesthetics or corticosteroids
* Patients with history of chronic pain or with chronic use of opioid analgesics
* Patients with history of lung disease or prior anterior thoracotomy or median sternotomy

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Alghoul, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.25 % Bupivacaine w/ Epinephrine & 4mg Dexamethasone: Subjects will be randomly selected to receive selective block with a local anesthetic solution containing 0.25 % bupivacaine (2.5 mg/ml) with 1:100,000 epinephrine and 4 mg dexamethasone. The injection will be performed in certain locations of the breast area to cover the intercostal nerves supplying the breast tissue.
  Subjects will be randomly selected to receive the local anesthetic solution containing 0.25 % bupivacaine (2.5 mg/ml) with 1:100,000 epinephrine and 4 mg dexamethasoneadministered to the breast area to cover the intercostal nerves supplying the breast tissue during surgery.
  0.25 % bupivacaine (2.5 mg/ml) w/ 1:100,000 epinephrine & 4 mg dexamethasone: If randomized to this arm, subjects will receive a selective block with a local anesthetic solution containing 0.25 % bupivacaine.
  (2.5 mg/ml) with 1:100,000 epinephrine and 4 mg dexamethasone intraoperatively.
Period: Overall Study
Arm/Group | Placebo | 0.25 % Bupivacaine w/ Epinephrine & 4mg Dexamethasone
Started | 23 | 24
Completed | 22 | 23
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.25 % Bupivacaine w/ Epinephrine & 4mg Dexamethasone | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [42 to 57] | 48 [43 to 58] | 49 [43 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery Score
Description: The primary outcome measure is a well-validated and widely used survey measuring the quality of recovery from anesthesia entitled the "Global 40 Item Quality of Recovery" survey. This is a 40 question survey administered to patients to allow them to rate their quality of recovery along a number of different dimensions, including emotional state, physical comfort, psychological support, physical independence, and pain. The score ranges from 40 to 200, with 40 representing a very poor overall quality of recovery and 200 representing the best possible recovery. The following reference explains the Global 40 Item Quality of Recovery survey in detail:
  Myles, P.S., et al., Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth, 2000. 84(1): p. 11-5.
  PMID: 10740540
Time Frame: 24 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | 0.25 % Bupivacaine w/ Epinephrine & 4mg Dexamethasone
Number analyzed (Participants) | 22 | 23
score on a scale | 165 [143 to 179] | 169 [155 to 182]

2. Secondary Outcome: Pain Score Using 10-point Visual Analog Scale (VAS)
Description: A study-specific pain form was provided to the patient and nursing staff that consisted of standard visual analogue scale (VAS) for patients to rate their pain level. Pain level was rated as a categorical level from 0 to 10, in 1 unit increments, with 0 being "no pain at all" and 10 being "worst pain imaginable." Thus a total of 10 pain grades were possible.
Time Frame: 24 hrs
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | 0.25 % Bupivacaine w/ Epinephrine & 4mg Dexamethasone
Number analyzed (Participants) | 22 | 23
score on a scale | 4 [2 to 6] | 4 [3 to 6]

3. Secondary Outcome: Opioid Consumption
Description: Total opioid consumption in the first 24 hrs of recovery after surgery as measured in "morphine equivalents." This involves converting the dose of a non-morphine narcotic (e.g. IV hydromorphone or oral hydrocodone) into the equi-analgesic dose of morphine, so that the total amount of narcotic utilized by the patient can be compared. This is a standard technique for comparison utilized in the pain management literature.
Time Frame: 24 hrs
Measure: Median (Inter-Quartile Range); unit: Morphine equivalents
Arm/Group | Placebo | 0.25 % Bupivacaine w/ Epinephrine & 4mg Dexamethasone
Number analyzed (Participants) | 22 | 23
Morphine equivalents | 114 [69 to 161] | 92 [44 to 142]

4. Secondary Outcome: Length of Hospital Stay
Description: Number of postoperative days patients stay in the hospital after surgery
Time Frame: 4 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | 0.25 % Bupivacaine w/ Epinephrine & 4mg Dexamethasone
Number analyzed (Participants) | 22 | 23
Days | 1 [1 to 1] | 1 [1 to 1]

ADVERSE EVENTS:
Arm/Group | Placebo | 0.25 % Bupivacaine w/ Epinephrine & 4mg Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes